CLINICAL TRIAL: NCT02060214
Title: Development of Novel Cystometrics for Overactive Bladder
Status: Withdrawn | Type: Observational
Why Stopped: Study unable to enroll due to feasibility issues
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20000453
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Urinary Frequency/Urgency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Urinary urgency is the key symptom of overactive bladder (OAB). A critical barrier in understanding OAB is the lack of a method to separate urgency that derives directly from bladder filling or what we term "tension sensor output" and urgency that derives from abnormal brain interpretation. The central hypothesis is that measureable biomechanical parameters can directly affect the output (urgency) of the detrusor tension sensor.

The development of novel cystometric tests for the improved diagnosis and treatment of OAB and for the potential identification of novel mechanistic targets in the pathophysiology of OAB.

DETAILED DESCRIPTION:
Aim 1. Validate an Urgency Meter and quantify urgency-volume relationship. Test the hypothesis that the tension sensor output of urinary urgency can be objectively measured and is reflected by the input of filling volume.

Aim 2. Quantify the bladder geometry-urgency relationship. Test the hypothesis that bladder geometry (wall thickness, surface area, and shape) affects the load on the detrusor tension sensor as reflected by objective changes in the output of urgency.

Aim 3. Quantify the dynamic compliance-urgency relationship. Test the hypothesis that dynamic compliance (strain-history and activation-history dependent compliance) affects the load on the detrusor tension sensor as reflected by objective changes in the output of urgency.

Aim 4. Quantify the spontaneous rhythmic contraction-urgency relationship. Test the hypothesis that spontaneous rhythmic contractions affect the load on the detrusor tension sensor as reflected by objective changes in the output of urgency.

Urinary urgency is the key symptom in Overactive Bladder (OAB) that occurs during the filling phase of micturition, and increased detrusor wall tension is thought to be a critical factor in the pathophysiology of OAB. However, because pressure increases little during bladder filling and does not reflect changes in detrusor wall tension, true filling phase physiology cannot be evaluated during clinical cystometrics. Thus, objective assessments of OAB using standard clinical cystometric testing is difficult or impossible. Furthermore, evaluation of OAB using verbal sensory thresholds recommended by the International Continence Society are subjective and poorly defined. Thus, there is a pressing need for a mechanistically relevant diagnostic test of OAB that incorporates objective metrics for the direct evaluation of detrusor wall tension.

Using a systems model of the filling phase of micturition, the detrusor smooth muscle and its in-series tension sensitive afferent nerves can be represented as a tension sensor with a definable input (volume), an objectively measurable output (urgency), and objectively measurable biomechanical parameters that affect the load on the tension sensor. Based on our previous investigations and the work of others, we have identified the following biomechanical parameters that can directly affect the load on the detrusor tension sensor during filling: bladder geometry, dynamic compliance, and spontaneous rhythmic contractions. In the current proposal, we will develop novel cystometric tests to assess bladder geometry, dynamic compliance, and spontaneous rhythmic contractions during the filling phase of micturition. Our new cystometrics will include 1) a sliding scale Urgency Meter that will allow patients to continuously record the tension sensor output of urgency, 2) two and three dimensional bladder ultrasonography to provide real-time measurements of bladder geometry that will be used to measure the effect of geometry and used for dynamic compliance calculations, and 3) Fast Fourier Transform (FFT) analysis to objectively measure filling phase spontaneous rhythmic contractions

These new metrics will provide a quantitative mechanistic link between OAB symptomatology and detrusor function, and we will use these new metrics to identify tension-mediated and non-tension mediated sub-groups of OAB. In this proposal, our central hypothesis, that measurable biomechanical parameters can directly affect the output (urgency) of the detrusor tension sensor, will be tested in clinical experiments involving accelerated hydration, abbreviated cystometrics, and repeat-fill cystometrics, and extended-hold cystometrics. Successful completion of this multi-PI proposal involving the combined skill sets of a neuro-urologist and a mechanical engineer will allow for the development of novel cystometric tests for the improved diagnosis and treatment of OAB and for the potential identification of novel mechanistic targets in the pathophysiology of OAB.

ELIGIBILITY:
Inclusion Criteria:

Study 1:

* Inclusion for Control Subjects:
* No urgency defined as scoring a "0" on the screening question 5A of ICIQ-OAB survey instrument.
* Above 21 years of age.
* Healthy enough to undergo testing
* No Cognitive Impairment
* No vulnerable population

Inclusion for Heightened Urgency Group:

* Answer greater than or equal to 3 on question 5a of ICIQ-OAB survey instrument.
* Above 21 years of age.
* Healthy enough to undergo testing.
* Have no cognitive impairment.
* Not vulnerable population

Study 2, 3 and 4:

* Scheduled to undergo cystoscopy examinations for clinically indicated condition.
* Over 21 years of age.
* No cognitive impairment.
* No vulnerable population

Exclusion Criteria:

Study 1:

Exclusion for Control Participants:

* Prescription medications.
* Significant medical conditions.
* 21 years of age or younger
* Cognitive impairment.
* Vulnerable population.
* Scoring anything other than "0" on all screening questions on the ICIQ-OAB.
* Score less than or equal to 3 on question 5a of ICIQ--OAB.

Exclusion for Heightened Urgency Group:

* Significant medical conditions.
* 21 years of age or younger.
* Cognitive impairment.
* Vulnerable population.
* Score less than 3 on question 5a of ICIQ-OAB.

Study 2, 3, and 4:

* Not undergoing standard of care cystoscopy examinations for clinically indicated conditions.
* 21 years of age or younger.
* Have cognitive impairment.
* Vulnerable population

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample and Urology Clinic Patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Overactive Bladder/Urgency | one year
  validating the use of a computer program which will assist patients in describing their level of urgency. This and the use of ultrasound measurements of the bladder will assist us in developing a means to measure urgency for normal, healthy participants and those with elevated urgency.

CONTACTS AND LOCATIONS:
Overall Officials: Adam P Klausner, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States